CLINICAL TRIAL: NCT02130245
Title: Acute Cholecystitis: Early Versus Delayed Laparoscopic Cholecystectomy; Randomized Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, PhD, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Early cholecystectomy
Record Dates: First submitted 2014-04-21; First posted 2014-05-05 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Acute Cholecystitis
Keywords: Laparoscopic cholecystectomy; Acute cholecystitis; Early; Delayed
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early cholecystectomy (Active Comparator): Laparoscopic cholecystectomy well be done after the immediate admission
  Interventions: Procedure: Early cholecystectomy
- Delayed cholecystectomy (Active Comparator): Laparoscopic cholecystectomy after a period of conservative treatment
  Interventions: Procedure: Delayed cholecystectomy

INTERVENTIONS:
Procedure: Early cholecystectomy — Early laparoscopic cholecystectomy for acute cholecystitis after admission
  Other Names: First group
  Arms: Early cholecystectomy
Procedure: Delayed cholecystectomy — Laparoscopic cholecystectomy well be done after a period on conservation
  Other Names: Second group
  Arms: Delayed cholecystectomy

SUMMARY:
The best management of the acute cholecystitis is to do laparoscopic cholecystectomy. The hypothesis is that to do it as an early intervention after patient admission is better than delayed cholecystectomy regarding the hospital stay, interval for antibiotic, the easiness of the operative maneuver reflected by operative time, conversion and intraoperative complications.

DETAILED DESCRIPTION:
Doing laparoscopic cholecystectomy for patients with acute cholecystitis as an early intervention after patient admission ( first group) or to do it after a while of treatment and conservation as a delayed cholecystectomy (second group) points of study include the hospital stay, interval for antibiotic, the easiness of the operative maneuver reflected by operative time, conversion and intraoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Proved acute cholecystitis clinical, radiologic

Exclusion Criteria:

* Evidence of peritonitis
* ASA III or IV
* Previous upper abdominal surgery
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | 1 DAY
  Operative time is assessed in minutes ,

SECONDARY OUTCOMES:
Perioperative complications | 5 weeks
  Intraoperative complications like bleeding , injury,
Conversion rate | 1 DAY
  Conversion rate from laparoscopic to open and reason of conversion.
hospital stay in days | 2 weeks
  hospital stay in days
Period of giving antibiotics in days | 2 WEEKS
  Number of days giving the antibiotics

CONTACTS AND LOCATIONS:
Locations (1):
- mansoura university hospital, EGYPT, central hafr elbatin hospital, Saudia Arabia, Al Mansurah, Egypt

REFERENCES:
- See also: Related Info — http://www.mans.edu.eg/en